CLINICAL TRIAL: NCT05412745
Title: Head-to-head, Randomized Pivotal Study to Evaluate the Effect of a Class I Pullulan Based Medical Device Containing Allium Cepa and Hyaluronic Acid Compared to Class I Medical Device Silicone Gel on Post-surgical Scars
Brief Title: Class I Medical Device on Post-surgical Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Elena Campione, Professor Elena Campione, University of Rome Tor Vergata
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R.S. 211.19
Record Dates: First submitted 2022-05-25; First posted 2022-06-09 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Cicatrix; Post-Surgical Complication; Scar Itching; Keloid; Hypertrophic Scar
Keywords: scar; Keloid; Cicatrix; allium cepa; silicone
MeSH Terms: conditions — Cicatrix; Keloid; Cicatrix, Hypertrophic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): class I pullulan based medical device containing Allium cepa & HA
  Interventions: Device: Kaloidon Plus
- Group B (Active Comparator): class I medical device silicone gel
  Interventions: Device: silicone gel

INTERVENTIONS:
Device: Kaloidon Plus — topical application; twice daily
  Arms: group A
Device: silicone gel — topical application; twice daily
  Arms: Group B

SUMMARY:
To compare the effect of a class I pullulan based medical device containing Allium cepa & HA versus a class I medical device silicone gel on new post-surgical wounds

DETAILED DESCRIPTION:
A head-to-head, randomised, pivotal controlled trial evaluating the appearance of post-surgical scars for 12 weeks. The study was developed in 10 months, including recruitment, evaluation every 4 weeks and evaluation of the secondary objective in the third month (T2). The primary endpoint was the evaluation of the effectiveness of the class I medical device contain onion (Allium cepa) extract compared to the silicone gel used in the treatment of post-surgical scars for the prevention of hypertrophic scars. Objective scar assessment using the Vancouver Scar Scale (VSS), Manchester Scale, Patient and Observer Scar Assessment Scale (POSAS), itching, redness and pliability were performed after 4,8 and 12 weeks of treatment. Safety was also evaluated by gathering adverse events related to application of the gel. The statistical analysis of the data was carried out by applying parametric or non-parametric tests depending on the distribution of the data that was going to be obtained. The one-way analysis of variance ANOVA test was used to evaluate the reduction/increase of clinical parameters in the pre-established observation times (T0, T2, T3 and T4) for each treatment, whereas comparison between treatments was performed via t-test analysis. Correlation tests were also used. The differences were considered statistically significant for p values <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 and 70 who have undergone surgery for the excision of skin lesions at least 20 days before the start of the protocol.

Exclusion Criteria:

* Subjects affected by spontaneous keloids

  * Diabetic subjects with a previous history of disorders in the repair of wounds;
  * Subjects with overinfected wounds after the first week after surgery;
  * Subjects with documented sensitivity to silicone gel;
  * Subjects affected by collagen disorders (e.g. Pseudoxantoma elasticum, poikilodermatosis).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-09-10 (Actual); Study Completion 2022-09-10 (Actual)

PRIMARY OUTCOMES:
Change of Vancouver Scar Scale (VSS) | week 4,8,12
  Change of Vancouver Scar Scale (VSS) from baseline to weeks 4,8 and 12.
  * vascularity(range from normal(0 point) to purple(3point)
  * pigmentation(range from normal(0 point) to hyper-pigmentation(3point)
  * pliability(range from normal(0 point) to contracture(5point)
  * height (range from flat(0 point) to above 5mm(3point)
  * pain(range from none(0 point) to Require medication(2point)
  * itchiness(range from none(0 point) to Require medication(2point) We assess total score that are minimum score is 0 and maximum is 18. The lowest score means the best scar condition.
Change of Manchester Scale | week 4,8,12
  Change of Manchester Scale from baseline to weeks 4,8 and 12.
  * Color (range from perfect (1 point) to Gross mismatch (4 points)
  * Shine ( from matte (1 point) to shiny (2 points))
  * Contour ( from Flush with surrounding skin (1 point) to keloid (4 points))
  * Distortion ( from none (1 point) to severe (4 points)) Lower score denotes a better outcome using the MSS (range: 4-14).
Change of Patient and Observer Scar Assessment Scale (POSAS) from baseline to weeks 4,8 and 12. | week 4,8,12
  Change of Patient and Observer Scar Assessment Scale (POSAS) from baseline to weeks 4,8 and 12. Lower score denotes a better outcome using the POSAS (range: 0-10).
Change of itching from baseline to weeks 4,8 and 12 | week 4,8,12
  Change of itching from baseline to weeks 4,8 and 12 will be measure with the visual analogue scale (VAS). Lower score denotes a better outcome using the VAS (range: 0-10).
Change of redness from baseline to weeks 4,8 and 12 | week 4,8,12
  Change of redness from baseline to weeks 4,8 and 12 will be evaluted as 10 points scale, from normal (1 point) to purple (10 points). Lower score denotes a better outcome (range: 0-10).
Change of pliability from baseline to weeks 4,8 and 12 | week 4,8,12
  Change of pliability from baseline to weeks 4,8 and 12 will be measured by testing folding of the scar with a six-step scale: normal, supple, yielding, firm, banding, and contracture. Lower score denotes a better outcome (range: 0-10).

SECONDARY OUTCOMES:
Incidence of adverse events occurrence after treatment | week 12
  Incidence of adverse events will be evaluated since the baseline visit until 12 weeks after the end of the treatment. Adverse Events reported by patients or noticed by investigator will be reported as local skin reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Campione, Principal Investigator — University of Rome Tor Vergata
Locations (2):
- Italy (2):
  - Elena Campione, Roma
  - Tor Vergata Univerisity Hospital, Rome

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cosio T, Costanza G, Coniglione F, Romeo A, Iacovelli F, Diluvio L, Dika E, Shumak RG, Rossi P, Bianchi L, Falconi M, Campione E. From In Silico Simulation between TGF-beta Receptors and Quercetin to Clinical Insight of a Medical Device Containing Allium cepa: Its Efficacy and Tolerability on Post-Surgical Scars. Life (Basel). 2023 Aug 21;13(8):1781. doi: 10.3390/life13081781. PMID 37629638